CLINICAL TRIAL: NCT05195866
Title: Using the CRP Test in Children Under 12 Years With Respiratory Symptoms in Kyrgyz Republic
Brief Title: CRP for Respiratory Diagnosis in Kyrgyz Pediatric Practice
Acronym: COORDINATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: National Center of Maternity and Childhood Care (Unknown); National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); The Research Unit for General Practice (Unknown); Copenhagen School of Global Health (Unknown); Unit of Global Health, The Juliane Marie Center, Rigshospitalet (Unknown); Kyrgyz Thoracic Society (Unknown)
Responsible Party: Principal Investigator, Jesper Kjærgaard, Coordinator, Global Health Unit, Department of Paediatrics and Adolescent Health, Principal Investigator, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRPKG
Record Dates: First submitted 2021-11-24; First posted 2022-01-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Antibiotic Resistance; Respiratory Tract Infections; Pediatric Infectious Disease; CRP
Keywords: antibiotic resistance; respiratory tract infections; crp; respiratory symptoms; acute respiratory tract infections; CRP POCT; Pediatrics
MeSH Terms: conditions — Respiratory Tract Infections; Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: Individually randomized clinical trial
  The children will be randomized into two groups. Randomization will be stratified by male/female as well as age <5 years and >5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - CRP POCT (Active Comparator): Participants assigned to Group A will take C-reactive protein (CRP) point of care test (POCT) during a check-up with their healthcare worker (HCW). The assistant investigator will attend the child's consultation with the local HCW and complete the case report form (CRF). Consequently, the CRP result will be recorded in the CRF, which will be the basis for choosing a treatment, depending on its result.
  Interventions: Diagnostic Test: CRP POCT (C-reactive protein point of care test)
- Group B - Usual care (No Intervention): HCWs will also consult children who have been randomised to Group B. The assistant investigator will complete the CRF for these children, but the CRP POCT will not test them. They will receive the treatment prescribed by the HCW as usual care

INTERVENTIONS:
Diagnostic Test: CRP POCT (C-reactive protein point of care test) — CRP POCT equipment will be supplied at healthcare centers, along with a short training in use and interpretation supporting the clinical evaluation of the child. It will be communicated that CRP levels less than 10 indicate that the disease is not severe, and antibiotics is most likely not needed, if between 10 and 50, that antibiotics might be needed, and if more than 50 that it is likely that they are needed. With CRP between 10-50 the HCW are instructed to take the clinical picture into account together with the value of the test.
  The training will also include knowledge of CRP pharmacodynamics and cases where a low CRP might need to be interpreted cautiously, e.g. a history of fever lasting less than 24 hrs. HCWs will be instructed to use CRP POCT for all patients in the intervention group and use the information to guide diagnosis and treatment choice. We will use Aidian (Copenhagen, Denmark) QuickRead go CRP POCT set-up.
  Arms: Group A - CRP POCT

SUMMARY:
Rationale:

Overuse of antibiotics globally is leading to increasing rates of antibiotic resistance and may lead to a 'post-antibiotic' era. Case fatality rates for pneumonia in children remain high in Central Asia and there is a lack of knowledge of which viruses and bacteria cause the disease. Antibiotic resistance patterns of common bacteria remain largely unknown in Central Asia which makes it challenging for clinicians to choose the right antibiotic to treat children with suspected bacterial pneumonia and sometimes healthcare workers overuse an antibacterial therapy even when the child does not need it.

Randomised trials of using CRP point of care test (POCT) to guide antibiotic prescription for respiratory tract infections has been successful in lowering unnecessary antibiotic prescriptions in adults in high income countries but left a small concern for safety in the form of possibly slightly increased risk of hospitalisation in the CRP group.

Objective:

This study seeks to gain evidence on whether use of C-reactive protein point-of-care test can safely decrease prescription of antibiotics for children under 12 with acute respiratory symptoms in primary level healthcare centres in Kyrgyzstan.

Study design:

Multicentre, open-label, individual randomised controlled clinical trial with 14 days blinded follow-up in rural Chui and Naryn regions of Kyrgyz Republic. Healthcare workers from ten selected healthcare centres will be trained in the CRP POCT and in interpreting the results in the field.

Study population:

Children aged from 6 month to 12 years attending the primary level healthcare centres during normal business hours with acute respiratory symptoms.

Main study parameters:

The proportion of patients in the two groups prescribed an antibiotic within 14 days of index consultation; length of disease, antibiotics given at index consultation, admissions and vital status.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Risks, inconvenience and burden associated with participating in this observational study are low. As part of the inclusion children in the CRP cluster group will have a finger-prick test performed. This may be unpleasant and course transient discomfort but poses no risks to the child. Follow-up will be three short phone calls day 3, 7 and 14 after inclusion. Risks includes possible undertreatment of serious disease, however previous studies have not found safety issues with CRP testing in children. There is no direct benefit to participants, but side effects and non-necessary medications are likely minimised.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Respiratory tract infections are the most common cause of contact to the health system and are the main reason for antibiotic overuse at the primary care level globally. At the same time, acute lower respiratory infections (ALRI) are the most common cause of death among children under 5 globally, costing the lives of almost 1 million children annually. Unfortunately, there is substantial overlap in the presentation of different causes of acute lower respiratory illness in young children, including bacterial pneumonia, viral infections and wheezing and with increasing coverage of pneumococcal and Haemophilus influenza type b vaccination, only a smaller proportion of these need antibiotics. At the same time, globally, most children are diagnosed and treated at a primary care clinic, primarily by mid-level providers with only limited access to diagnostic equipment. To assist healthcare providers in diagnosing under these conditions, various algorithms have been used, e.g. WHO's Integrated Management of Childhood Illness, which bases diagnosis of respiratory diseases in children mainly on presence of cough and elevated respiratory rate. This approach has been shown to severely over-diagnose pneumonia and thus result in unnecessary prescription of antibiotics. Therefore, new approaches to diagnosing and treating respiratory infections in children are urgently needed.

Concurrently, antimicrobial resistance is now what WHO calls a global health emergency and warns that 'A post-antibiotic era - in which common infections and minor injuries can kill - far from being an apocalyptic fantasy, is instead a very real possibility for the 21st century. Unnecessary prescription of antibiotics is extensive globally and most healthcare providers are aware of the global threat of antimicrobial resistance but express the need for support for prescribing differently, such as knowledge of local resistance patterns of pathogens and better diagnostics to support a decision not to treat with an antibiotic.

C-reactive protein (CRP) is an acute phase reactant produced by the liver which can be used as a marker of serious infection. Randomised trials of using CRP point of care test (POCT) to guide antibiotic prescription for respiratory tract infections has been successful in lowering unnecessary antibiotic prescriptions in adults in high income countries but left a small concern for safety in the form of possibly slightly increased risk of hospitalisation in the CRP group. Trials of CRP POCT in children have been performed in Tanzania as part of an intervention package with a strict prescription limit of > 80 mg/L CRP with a reduction in antibiotic prescriptions from 40% to 2%. In South-East Asia with a small but statistically significant effect (5% reduction) when used as either above or below a certain threshold (40 mg/L) in Thailand and Myanmar. In a sub-group analysis from a trial in Vietnam with both children and adults where the numeric value of CRP was used after a short training in CRP interpretation along with clinical evaluation resulted in a 20% reduction from 64% to 44%. A cross-cutting qualitative study of the above-mentioned studies in Thailand, Myanmar, and Vietnam showed that lack of non-antibiotic alternatives to prescribe led to lower adherence to the CRP POCT result.

As the intervention of supplying CRP POCT to healthcare providers is more a behavioural than biomedical, previous trials have recommended that further trials are done in different contexts and that qualitative studies of reasons for success or failure.

Central Asian countries have been underrepresented in health science, especially in primary care research. The clinical context of primary care in South-East Asian countries, like Vietnam, Thailand, and Myanmar, and Central-Asian countries, like Kyrgyzstan, are vastly different with different caseloads, different human resources, and varying time for consultations available. At the same time, case fatality rates for pneumonia in children remain high in Central Asia and there is a lack of knowledge of which viruses and bacteria cause the disease. Antibiotic resistance patterns of common bacteria remain largely unknown in Central Asia, which makes it challenging for clinicians to choose the right antibiotic to treat children with suspected bacterial pneumonia. Kyrgyz Republic with respiratory diseases being the most common (49,7%). Among all acute respiratory diseases in children, upper respiratory tract infections are the most common. The number of cases per 100,000 population seems to de-crease by 2020, but it is still quite high.

OBJECTIVES

The aim of this project is to find out if the overuse of antibiotics in children with acute respiratory symptoms can be reduced by effectively identifying children at increased risk of infections who require antibiotic therapy and children who will not benefit from antibiotics. This is done by implementing CRP POCT at the primary healthcare level.

Hypotheses:

Supplying CRP POCT equipment to primary healthcare providers will help them identify the majority of children who suffer from viral infections and assist in withholding antibiotic treatment when no benefit can be expected and will help identify the severely sick children in need of urgent referral, thus lowering unnecessary use of antibiotics and improving primary care management by studying supplying supportive medication for those not in need of antibiotics.

It will be an individually randomised clinical trial where CRP POCT is supplied to approximately 14 healthcare centres. All children up to 12 years with respiratory symptoms have basic clinical data recorded as well as data needed to classify according to WHO IMCI pneumonia diagnostic criteria. CRP POCT is used at intervention sites and CRP results, diagnosis, and treatment is recorded. Follow-up phone calls will be made 3, 7 and 14 days after the health centre visit to record recovery, antibiotics use, hospitalisation and vital status of the participating children.

Ethics and dissemination: The study was approved 25/06/2021 by National center of Maternity and Childhood Care Ethics Committee (ref: no. 1). Study results will be disseminated through appropriate peer-reviewed journals, national and international respiratory conferences, social media, and through patient and public involvement events in Kyrgyzstan and in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 month and 12 years of age;
* Parents/caregivers of a child are able and willing to comply with all study requirements;
* Parents/caregivers of a child is able and willing to give Informed Consent;
* Having at least one of the following focal symptoms lasting for less than 2 weeks (cough; fast/difficult breathing; dore throat; shortness of breath; wheezing)

Exclusion Criteria:

* Severely ill and in need of urgent referral where measurement of CRP POCT would delay the process;
* Terminally ill patients;
* Patients with ear ache only;
* Patients with known immunosuppression or severe chronic disease (HIV, liver disease, history of neoplastic disease, long term systemic steroid use or similar conditions as assessed by the health worker or AI);
* Parents/caregivers who are not able to participate in follow-up procedures (lack of telephone etc);
* Haven taken antibiotics within 24 hours before the index consultation

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1204 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Proportion of children receiving antibiotics | Up to 1 year
  The primary study outcome is the proportion of included children in each study arm that are prescribed an antibiotic within 14 days from the index consultation (superiority analysis).
Patient safety | Up to 1 year
  The second primary study outcome is patient safety measured as the number of days until recovery (non-inferiority analysis).

SECONDARY OUTCOMES:
Antibiotics prescribed at the index consultation | Up to 1 year
  Number of children who were prescribed antibiotics at the index consultation
Antiviral treatment at follow up | Up to 1 year
  Number of children who were prescribed antiviral treatment at the follow up
Reconsultation within 14 days from index consultation | Up to 1 year
  Number of reconsultations within 14 days from index consultation
Hospital referral at index consultation | Up to 1 year
  Number of hospitalisations at index consultation
Hospital admission at follow up | Up to 1 year
  Number of hospital admissions at follow up
Mortality | Up to 1 year
  Number of children who died from the index consultation till the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Kjærgaard, MD, PhD, Study Chair — Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark; Elvira Isaeva, Dr., Principal Investigator — National Center of Maternity and Childhood Care, Bishkek, Kyrgyzstan; Talant Sooronbaev, MD, Professor, Study Director — Republican Research Centre of Pulmonology and Rehabilitation the Ministry of Health of the Kyrgyz Republic
Locations (1):
- At-Bashy FMC, Naryn, Naryn Region, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aabenhus R, Jensen JU, Jorgensen KJ, Hrobjartsson A, Bjerrum L. Biomarkers as point-of-care tests to guide prescription of antibiotics in patients with acute respiratory infections in primary care. Cochrane Database Syst Rev. 2014 Nov 6;(11):CD010130. doi: 10.1002/14651858.CD010130.pub2. PMID 25374293
- [Background] Risk R, Naismith H, Burnett A, Moore SE, Cham M, Unger S. Rational prescribing in paediatrics in a resource-limited setting. Arch Dis Child. 2013 Jul;98(7):503-9. doi: 10.1136/archdischild-2012-302987. Epub 2013 May 9. PMID 23661572
- [Background] Havers FP, Hicks LA, Chung JR, Gaglani M, Murthy K, Zimmerman RK, Jackson LA, Petrie JG, McLean HQ, Nowalk MP, Jackson ML, Monto AS, Belongia EA, Flannery B, Fry AM. Outpatient Antibiotic Prescribing for Acute Respiratory Infections During Influenza Seasons. JAMA Netw Open. 2018 Jun 1;1(2):e180243. doi: 10.1001/jamanetworkopen.2018.0243. PMID 30646067
- [Background] Kjaergaard J, Anastasaki M, Stubbe Ostergaard M, Isaeva E, Akylbekov A, Nguyen NQ, Reventlow S, Lionis C, Sooronbaev T, Pham LA, Nantanda R, Stout JW, Poulsen A; FRESH AIR Collaborators. Diagnosis and treatment of acute respiratory illness in children under five in primary care in low-, middle-, and high-income countries: A descriptive FRESH AIR study. PLoS One. 2019 Nov 6;14(11):e0221389. doi: 10.1371/journal.pone.0221389. eCollection 2019. PMID 31693667
- [Background] Hug L, Sharrow D, You D. Levels & Trends in Child Mortality. New York, 2017 http://www.childmortality.org/files_v21/download/IGME report 2017 child mortality final.pdf.
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Zar HJ, Ferkol TW. The global burden of respiratory disease-impact on child health. Pediatr Pulmonol. 2014 May;49(5):430-4. doi: 10.1002/ppul.23030. Epub 2014 Mar 9. PMID 24610581
- [Background] Lai CK, Beasley R, Crane J, Foliaki S, Shah J, Weiland S; International Study of Asthma and Allergies in Childhood Phase Three Study Group. Global variation in the prevalence and severity of asthma symptoms: phase three of the International Study of Asthma and Allergies in Childhood (ISAAC). Thorax. 2009 Jun;64(6):476-83. doi: 10.1136/thx.2008.106609. Epub 2009 Feb 22. PMID 19237391
- [Background] Hazir T, Nisar YB, Abbasi S, Ashraf YP, Khurshid J, Tariq P, Asghar R, Murtaza A, Masood T, Maqbool S. Comparison of oral amoxicillin with placebo for the treatment of world health organization-defined nonsevere pneumonia in children aged 2-59 months: a multicenter, double-blind, randomized, placebo-controlled trial in pakistan. Clin Infect Dis. 2011 Feb 1;52(3):293-300. doi: 10.1093/cid/ciq142. Epub 2010 Dec 28. PMID 21189270
- [Background] Shao AF, Rambaud-Althaus C, Samaka J, Faustine AF, Perri-Moore S, Swai N, Kahama-Maro J, Mitchell M, Genton B, D'Acremont V. New Algorithm for Managing Childhood Illness Using Mobile Technology (ALMANACH): A Controlled Non-Inferiority Study on Clinical Outcome and Antibiotic Use in Tanzania. PLoS One. 2015 Jul 10;10(7):e0132316. doi: 10.1371/journal.pone.0132316. eCollection 2015. PMID 26161535
- [Background] WHO. Integrated Management of Childhood Illness Chart Booklet. 2014.
- [Background] Nantanda R, Tumwine JK, Ndeezi G, Ostergaard MS. Asthma and pneumonia among children less than five years with acute respiratory symptoms in Mulago Hospital, Uganda: evidence of under-diagnosis of asthma. PLoS One. 2013 Nov 29;8(11):e81562. doi: 10.1371/journal.pone.0081562. eCollection 2013. PMID 24312321
- [Background] WHO. ANTIMICROBIAL RESISTANCE Global Report on Surveillance. Geneva, 2014 http://apps.who.int/iris/bitstream/10665/112642/1/9789241564748_eng.pdf?ua=1.
- [Background] O'Neill J. Tackling Drug-Resistant Infections Globally: Final Report and Recommendations. 2016 https://amr-review.org/sites/default/files/160525_Final paper_with cover.pdf.
- [Background] Keitel K, Samaka J, Masimba J, Temba H, Said Z, Kagoro F, Mlaganile T, Sangu W, Genton B, D'Acremont V. Safety and Efficacy of C-reactive Protein-guided Antibiotic Use to Treat Acute Respiratory Infections in Tanzanian Children: A Planned Subgroup Analysis of a Randomized Controlled Noninferiority Trial Evaluating a Novel Electronic Clinical Decision Algorithm (ePOCT). Clin Infect Dis. 2019 Nov 13;69(11):1926-1934. doi: 10.1093/cid/ciz080. PMID 30715250
- [Background] Althaus T, Greer RC, Swe MMM, Cohen J, Tun NN, Heaton J, Nedsuwan S, Intralawan D, Sumpradit N, Dittrich S, Doran Z, Waithira N, Thu HM, Win H, Thaipadungpanit J, Srilohasin P, Mukaka M, Smit PW, Charoenboon EN, Haenssgen MJ, Wangrangsimakul T, Blacksell S, Limmathurotsakul D, Day N, Smithuis F, Lubell Y. Effect of point-of-care C-reactive protein testing on antibiotic prescription in febrile patients attending primary care in Thailand and Myanmar: an open-label, randomised, controlled trial. Lancet Glob Health. 2019 Jan;7(1):e119-e131. doi: 10.1016/S2214-109X(18)30444-3. PMID 30554748
- [Background] Do NT, Ta NT, Tran NT, Than HM, Vu BT, Hoang LB, van Doorn HR, Vu DT, Cals JW, Chandna A, Lubell Y, Nadjm B, Thwaites G, Wolbers M, Nguyen KV, Wertheim HF. Point-of-care C-reactive protein testing to reduce inappropriate use of antibiotics for non-severe acute respiratory infections in Vietnamese primary health care: a randomised controlled trial. Lancet Glob Health. 2016 Sep;4(9):e633-41. doi: 10.1016/S2214-109X(16)30142-5. Epub 2016 Aug 3. PMID 27495137
- [Background] Haenssgen MJ, Charoenboon N, Do NTT, Althaus T, Khine Zaw Y, Wertheim HFL, Lubell Y. How context can impact clinical trials: a multi-country qualitative case study comparison of diagnostic biomarker test interventions. Trials. 2019 Feb 8;20(1):111. doi: 10.1186/s13063-019-3215-9. PMID 30736818
- [Derived] Isaeva E, Bloch J, Akylbekov A, Skov RL, Poulsen A, Kurtzhals JAL, Reventlow S, Sreenivasan N, Mademilov M, Siersma VD, Sooronbaev T, Kjaergaard J, Aabenhus RM. C-reactive protein testing in primary care and antibiotic use in children with acute respiratory tract infections in Kyrgyzstan: an open-label, individually randomised, controlled trial. Lancet Reg Health Eur. 2025 Jan 10;51:101184. doi: 10.1016/j.lanepe.2024.101184. eCollection 2025 Apr. PMID 39886015
- [Derived] Isaeva E, Akylbekov A, Bloch J, Poulsen A, Kurtzhals J, Siersma V, Sooronbaev T, Aabenhus RM, Kjaergaard J. The Feasibility of C-Reactive Protein Point-of-Care Testing to Reduce Overuse of Antibiotics in Children with Acute Respiratory Tract Infections in Rural Kyrgyzstan: A Pilot Study. Pediatric Health Med Ther. 2024 Feb 13;15:67-76. doi: 10.2147/PHMT.S425095. eCollection 2024. PMID 38371485
- [Derived] Isaeva E, Bloch J, Poulsen A, Kurtzhals J, Reventlow S, Siersma V, Akylbekov A, Sooronbaev T, Munck Aabenhus R, Kjaergaard J. C reactive protein-guided prescription of antibiotics for children under 12 years with respiratory symptoms in Kyrgyzstan: protocol for a randomised controlled clinical trial with 14 days follow-up. BMJ Open. 2023 Apr 11;13(4):e066806. doi: 10.1136/bmjopen-2022-066806. PMID 37041063
- See also: CRP POCT — https://www.aidian.eu/point-of-care/quikread-go/quikread-go-easy-crp
- See also: SealedEnvelope Randomisation Programme — https://www.sealedenvelope.com/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT05195866/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT05195866/ICF_003.pdf